CLINICAL TRIAL: NCT06176755
Title: Effects of Treadmill Training With and Without Weighted Ankle Cuffs on Gait Parameters in Children With Down's Syndrome
Brief Title: Treadmill Training With and Without Weighted Ankle Cuffs on Gait Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: REC/RCR&AHS/23/0749
Record Dates: First submitted 2023-11-09; First posted 2023-12-20 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Down's Syndrome
Keywords: Berg Balance scale, Down syndrome, Gait parameter, Posture
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: Randomised Control Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treadmill training with weighted ankle cuffs (Experimental): Participants in group A will provided with small, motorized, custom-designed treadmills and trained parents to appropriately administer training in their homes. Parents held their infant upright on the treadmill at the front of the belt. The belt of the treadmill, when turned on, moved the infants' legs backward and elicited forward stepping. Whenever infants did not generate steps, parents repositioned the infant to the front of the belt. Infants will receive the protocol about 4 days a week for 1 hour/day for total of 6 weeks at a belt speed of 0.18m/sec. Besides progressively increasing belt speed and daily training duration, we attached to the infants' ankles a small amount of weight that was proportional to their estimated calf mass, and increased the weight over the course of training. Treadmill training terminated when participants walked three steps independently
  Interventions: Other: Treadmill training with weighted ankle cuffs
- Treadmill training (Active Comparator): Participants in group A will provided with small, motorized, custom-designed treadmills and trained parents to appropriately administer training in their homes. Parents held their infant upright on the treadmill at the front of the belt. The belt of the treadmill, when turned on, moved the infants' legs backward and elicited forward stepping. Whenever infants did not generate steps, parents repositioned the infant to the front of the belt. Infants will receive the protocol about 4 days a week for 1 hour/day for total of 6 weeks at a belt speed of 0.18m/sec. Besides progressively increasing belt speed and daily training duration, we attached to the infants' ankles a small amount of weight that was proportional to their estimated calf mass, and increased the weight over the course of training. Treadmill training terminated when participants walked three steps independently.
  Interventions: Other: Treadmill training

INTERVENTIONS:
Other: Treadmill training with weighted ankle cuffs — Group A: Treadmill training and Ankle cuff.
  Participants in group A will provided with small, motorized, custom-designed treadmills and trained parents to appropriately administer training in their homes. Parents held their infant upright on the treadmill at the front of the belt. The belt of the treadmill, when turned on, moved the infants' legs backward and elicited forward stepping. Whenever infants did not generate steps, parents repositioned the infant to the front of the belt. Infants will receive the protocol about 4 days a week for 1 hour/day for total of 6 weeks at a belt speed of 0.18m/sec. Besides progressively increasing belt speed and daily training duration, we attached to the infants' ankles a small amount of weight that was proportional to their estimated calf mass, and increased the weight over the course of training. Treadmill training terminated when participants walked three steps independently.
  Arms: Treadmill training with weighted ankle cuffs
Other: Treadmill training — Treadmill training only
  Arms: Treadmill training

SUMMARY:
Down syndrome is a condition in which a person has an extra chromosome. Chromosomes are small "packages" of genes in the body. Down syndrome (DS), also known as trisomy 21, is caused by the presence of all or part of a third copy of chromosome 21. It is named after John Langdon Down, the British physician who described the syndrome for the first time in 1866.Down syndrome remains the most common chromosomal condition diagnosed in the United States.

Current study will be randomized controlled trial. Study will be approved by ethical committee. After that informed consent will be taken and patients will be included in the study based on the inclusion criteria. Sampling technique will be simple random sampling the calculated sample sizes will be 25 in each group. All participants will be divided in two groups. One group will receive treadmill training with Weighted Ankle Cuffs and second group will receive treadmill training only. Conventional therapy will be given to both groups which include isometric, strengthening exercise and trunk exercise. The exercise was given for 10 repetitions/session. Infants will receive the treadmill training protocol about 6 min/day, 4 day/week at a belt speed of 0.18m/sec. After taking informed consent baseline measurement will be taken through gait assessment rating scale and Berg balance scale for balance and Gait parameters respectively. Data will be collected before treatment and after 6 weeks. Treatment session will be performed for 1 hour per day, 4 days a week for total of 6 weeks. The difference in improvement before and after 4th weeks will be noted and compared through SPSS 26.0.

DETAILED DESCRIPTION:
Participants will complete a well-tested Performa. Gait parameters will be collected through these questions. The difference in improvement before and after 6th weeks will be noted and compared. Children receive treatment for 4 days a week for 1/day hour for total of 6 weeks.

Group A: Treadmill training and Ankle cuff.

Treadmill training:

Participants in group A will provided with small, motorized, custom-designed treadmills and trained parents to appropriately administer training in their homes. Parents held their infant upright on the treadmill at the front of the belt. The belt of the treadmill, when turned on, moved the infants' legs backward and elicited forward stepping. Whenever infants did not generate steps, parents repositioned the infant to the front of the belt. Infants will receive the protocol about 4 days a week for 1 hour/day for total of 6 weeks at a belt speed of 0.18m/sec. Besides progressively increasing belt speed and daily training duration, we attached to the infants' ankles a small amount of weight that was proportional to their estimated calf mass, and increased the weight over the course of training. Treadmill training terminated when participants walked three steps independently(18).

Weighted Ankle Cuffs: Choose the weight range. Wrap the weight cuff (0.5 kg) around the ankle, tighten enough to avoid sliding along the leg during exercise. Apply hook and loop closure for secured fit. Do change the weight as per advice given by your consultant.

Group B: Treadmill training only. Participants in group A will provided with small, motorized, custom-designed treadmills and trained parents to appropriately administer training in their homes. Parents held their infant upright on the treadmill at the front of the belt. The belt of the treadmill, when turned on, moved the infants' legs backward and elicited forward stepping. Whenever infants did not generate steps, parents repositioned the infant to the front of the belt. Infants will receive the protocol about 4 days a week for 1 hour/day for total of 6 weeks at a belt speed of 0.18m/sec. Besides progressively increasing belt speed and daily training duration, we attached to the infants' ankles a small amount of weight that was proportional to their estimated calf mass, and increased the weight over the course of training. Treadmill training terminated when participants walked three steps independently.

Children will receive treatment for 4 days a week for 1 hour/day for total of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age from 5 to 10 years
* Absence of visual and cognitive problems
* Level 1,2 or 3 on gross motor function scale
* Function ambulation for at least 12 months

Exclusion Criteria:

* Children submitted to orthopedic surgical procedures or neuromuscular block in the 12 Months prior to the training sessions
* those with orthopedic deformity with indication for surgery

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Berg balance scale for functional balance | 4weeks
  The Berg balance test - or Berg balance scale (BBS) - is a widely used assessment to determine a person's balance abilities(15). The test contains 14 simple tasks and the entire process takes about 20 minutes to complete. The absolute reliability of the Berg Balance Scale varies across the scale, with minimal detectable change with 95% confidence varying between 2.8/56 and 6.6/56. The absolute reliability is stronger at the high end and weaker towards the middle of the scale.
Gait Abnormality Rating Scale (GARS) | 4weeks
  Gait Abnormality Rating Scale (GARS) is a videotape-based analysis of 16 facets of human gait. It has been evaluated as a screening tool to identify patients at risk for injury from falls. and has been used in remote gait evaluation. A modified version was published in 1996

CONTACTS AND LOCATIONS:
Overall Officials: Asma Iqbal, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah international university, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] VanSwearingen JM, Paschal KA, Bonino P, Yang JF. The modified Gait Abnormality Rating Scale for recognizing the risk of recurrent falls in community-dwelling elderly adults. Phys Ther. 1996 Sep;76(9):994-1002. doi: 10.1093/ptj/76.9.994. PMID 8790277